CLINICAL TRIAL: NCT04322799
Title: A Randomized Controlled RSA Study Comparing the 2nd Generation Highly Cross-linked Polyethylene to Conventional Polyethylene in Cemented Total Hip Arthroplasty
Brief Title: A Randomized RSA Study Comparing HXLPE to Conventional Polyethylene in Cemented Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Kjell G Nilsson, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PolyvsHXLPE
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Hip; Arthroplasty Complications
Keywords: osteoarthritis; total hip arthroplasty; migration; wear
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: Two different acetabular cups in total hip arthroplasty. No difference in surgical surgical technique and type of stem. The cup have the identical outlining.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetabular cup HXLPE (Intervention) (Experimental): Randomization to HXLPE acetabular component.
  Interventions: Procedure: Device: Randomization between prosthetic components
- Acetabular cup Conventional PE (control) (Experimental): Randomization to Coventional PE as control group
  Interventions: Procedure: Device: Randomization between prosthetic components

INTERVENTIONS:
Procedure: Device: Randomization between prosthetic components — Patients are randomized between two types of cup components in total hip arthroplasty. Identical cups made of either highly-crosslinked polyethylene or conventional polyethylene.

SUMMARY:
A prospective randomized study comparing two types of cemented acetabular components, a highly-crosslinked polyethylene or conventional polyethylene in total hip arthroplasty. Primary outcome are component wear measured by RSA, secondary outcomes are migration and complications. Patients are evaluated 5 years postoperatively.

DETAILED DESCRIPTION:
Background:

Total hip replacements is a cost effective treatment of a symptomatic degenerative hip disease. Cemented total hip replacements are the most common implants in Sweden (Swedish hip registry, 2009).

Wear of ultra high molecular weight polyethylene has been a issue with regard to implant survival. At the time of the shift of the millennium highly cross-linked polyethylene was introduced to the markets. Experimental studies had shown reduction of wear in hip simulator studies (McKellop,1999). Subsequently the intention is to reduce osteolysis and implant loosening. Single surgeon pilot studies in the 1970 (Wroblevski et al. 1996, Oonishi 1998, Grobelaar 1999) were the first clinical series with good results leading to the development of 2nd generation highly cross-linked polyethylenes which is now the almost exclusively used PE worldwide. So far medium term clinical evaluation and laboratory assessment have showed reduced wear and good mechanical properties (Digas et al. 2003, 2004, 2007, Röhrl et al. 2005, 2007, D´Antonio et al. 2005)

Production of highly crosslinked polyethylene (HXLPE) consists of several steps. First the PE material is crosslinked by being subjected to either gamma irradiation of various intensity or electron beam irradiation. The second step is to remove the free radicals created during the irradiation. This is done either by annealing (i.e. warming up the PE to just under its melting temperature) or melting (i.e. warming up the PE to above its melting temperature). Finally, the implant is sterilized either by gamma irradiation or Ethylene Oxide and packed in vacuum or inert atmosphere.There are some possible drawbacks and challenges in the process of cross-linking polyethylene with regard to preserving the mechanical properties and elimination of free radicals (Kurtz et al. 2006, Currier et al. 2007).

Submelt annealing preserves mechanical properties but on the other hand cannot eliminate all free radicals existing in the PE. Retrieval-studies of some 2nd generation highly cross-linked polyethylenes manufactured in this way have shown signs of oxidation. The in-vivo oxidation has been located in the non articulating area such as the circumference of the acetabular liner. It has been discussed that the femoral head may protect the polyethylene against oxidation, and hence prevent the possible negative consequences of remaining free radicals (Currier et al 2007).

Melting the polyethylene eliminates all free radicals but alters the mechanical properties. This has led to PE cracks and implant failure in some clinical studies (Furmanski et al. 2009), whereas it has not been seen in other.

Finally, wear particles of highly crosslinked polyethylene are more often in the submicron size compared to conventional PE. Although these particles have a higher biological activity (Fisher et al. 2006), results of recent studies show however, that the overall risk for osteolysis and aggressiveness of highly cross-linked particles is reduced (Galvin et al. 2007).

Because of differences in the manufacturing processes of highly crosslinking PE between manufacturers (i.e. different GUR used, type of irradiation, intensity of irradiation, postirradiative treatment, type of sterilization and packing, etc, etc) all highly crosslinked polyethylenes differ somewhat from each other. One can not extrapolate results of in vitro or in vivo wear studies of one manufacturer to another. Also, because of these manufacturing differences, fixation characteristics may differ between the various types of HXLPEs. Therefore it is imperative that all new highly crosslinked polyethylenes are subjected to clinical studies of their wear and fixation performance using high accuracy methods before being used extensively.

Methods:

A prospective randomized study comparing acetabular components made of HXLPE or conventional PE in total hip arthroplasty. The study will be conducted at Department of Orthopaedics, Umeå University, Umeå, Sweden.

Aim of study The aim of the study is to compare the wear and migration of a 2nd generation polyethylene from Link with conventional polyethylene in an all-poly cemented acetabular cup of the Lubinus brand using radiostereometric analysis (RSA) with 5-year follow-up.

Hypothesis The H0-hypothesis is that the difference with in wear between HXLPE and conventional PE will not increase up to 5-year follow-up.

Material Patients (age 50 years and above) with primary osteoarthritis between 2013 and 2014 at the orthopaedic department at the county hospital (Lycksele) affiliated to Umeå University hospital, Sweden. Patients were treated with a cemented total hip arthroplasty. At surgery, after the acetabulum was reamed, randomization was performed by opening of a consecutively numbered sealed envelope informing whether a cup made of HXLPE or conventional PE should be inserted. The envelopes were kept far away from the operation theatre and were opened by a research nurse contacted by telephone. Randomization was stratified for gender. Within each stratum there was block randomization with 6 permutations in each block.

Patients have been followed for 5 years postoperatively.

Implants • Acetabular cup Intervention: Link-Ticona GUR 1020 HXLPE, 32 mm inner diameter (Trade name Lubinus® X-LINKed® )

Control: Link-Chirulene GUR 1020 UHMWPE, 32 mm inner diameter (Trade name Lubinus ® UHMWPE)

• Femur stem Test and control: Lubinus® SP II®, CrCo femoral head, 32 mm diameter

Radio Sterometric Analysis (RSA) Radiostereometric analysis measurements will be performed 5 years postoperatively.

Wear will be measured as penetration of the femoral head into the polyethylene in the proximal, proximo-medial (2D pm), proximo-posterior (2D pp), and proximo-medial-posterior (3D) directions. Since the penetration during the initial 3 months represents polyethylene yield or bedding in, wear measurements will be reported from 3 months and up to 5 years postoperatively.

Quality of cup fixation will be measured as rotations of the cup around the three cardinal axes in relation to acetabulum with the postoperative examination as reference.

The RSA measurements will be analysed at Umeå University Hospital. Patient data will be saved in a specific research database at Umeå University Hospital following specific guidelines from the national data security committee.

Ethical approval The study has been approved by the Ethics Committee of Umeå University (Dnr 2011-173-31M, 2018-34-31M).

Sample size With a mean difference in wear at 2 years of 0.1 mm or more (SD ± 0.1) between the groups (p< 0.05), 25 patients in each group will give a power of > 80%. In order to cater for losses during the follow up a total of 57 patients will be enrolled.

Scientific Value All new materials should be monitored closely and introduced in small study groups using a high precision measurement technique. Many markets require such tests before acceptance for general use is given. The new highly crosslinked polyethylene from Link-Ticona is not equivalent to current highly crosslinked polyethylenes on the market, and one can not extrapolate wear results from these other designs.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis
* Age 50 years and above
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up

Exclusion Criteria:

* Rheumatoid Arthritis
* Grossly abnormal hip anatomy (severe dysplasia)
* Fracture sequelae
* Patients who, as judged by the surgeon, are mentally incompetent or are reasonable unlikely to be compliant with the requirements of the study
* Immune suppression or grave systemic illness

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-02-07 (Actual); Primary Completion 2014-12-04 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Magnitude of Polyethylene Wear | 0-5 years
  The size of the femoral component penetration into the polyethylene measured in millimeters per year and the volumetric annual wear millimetres with radiostereometric (RSA) analysis of radiographs.

SECONDARY OUTCOMES:
Magnitude of Cup Migration | 0-5 years
  Migration measured in millimetres per year with radiostereometric (RSA) analysis of radiographs. Radiostereometric analysis (RSA) is a stereo X-ray technique used in clinical research studies to evaluate micro-motion and wear of orthopaedic implants within bone. The method has a high accuracy and precision. Technical requirements include the need for implanted marker beads and radiograph view angles determined by a calibration cage.
Surgical complications | 0-5 years
  Surgical complications and reapportions during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Nilsson, Professor, Principal Investigator — Umeå University
Locations (1):
- Lycksele hospital, Lycksele, Sweden

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: CSR
Time Frame: Publication at 1 year after completion of the study during 2020.
Access Criteria: International scientific peer-reviewed journal

REFERENCES:
- [Background] Digas G, Karrholm J, Thanner J, Herberts P. 5-year experience of highly cross-linked polyethylene in cemented and uncemented sockets: two randomized studies using radiostereometric analysis. Acta Orthop. 2007 Dec;78(6):746-54. doi: 10.1080/17453670710014518. PMID 18236180
- [Background] D'Antonio JA, Manley MT, Capello WN, Bierbaum BE, Ramakrishnan R, Naughton M, Sutton K. Five-year experience with Crossfire highly cross-linked polyethylene. Clin Orthop Relat Res. 2005 Dec;441:143-50. doi: 10.1097/00003086-200512000-00024. PMID 16330997
- [Background] Rajadhyaksha AD, Brotea C, Cheung Y, Kuhn C, Ramakrishnan R, Zelicof SB. Five-year comparative study of highly cross-linked (crossfire) and traditional polyethylene. J Arthroplasty. 2009 Feb;24(2):161-7. doi: 10.1016/j.arth.2007.09.015. Epub 2008 Mar 4. PMID 18534491
- [Background] Kurtz SM, Hozack WJ, Purtill JJ, Marcolongo M, Kraay MJ, Goldberg VM, Sharkey PF, Parvizi J, Rimnac CM, Edidin AA. 2006 Otto Aufranc Award Paper: significance of in vivo degradation for polyethylene in total hip arthroplasty. Clin Orthop Relat Res. 2006 Dec;453:47-57. doi: 10.1097/01.blo.0000246547.18187.0b. PMID 17031310
- [Background] Rohrl SM, Li MG, Nilsson KG, Nivbrant B. Very low wear of non-remelted highly cross-linked polyethylene cups: an RSA study lasting up to 6 years. Acta Orthop. 2007 Dec;78(6):739-45. doi: 10.1080/17453670710014509. PMID 18236179
- [Background] McKellop H, Shen FW, Lu B, Campbell P, Salovey R. Development of an extremely wear-resistant ultra high molecular weight polyethylene for total hip replacements. J Orthop Res. 1999 Mar;17(2):157-67. doi: 10.1002/jor.1100170203. PMID 10221831
- [Background] Lerf R, Zurbrugg D, Delfosse D. Use of vitamin E to protect cross-linked UHMWPE from oxidation. Biomaterials. 2010 May;31(13):3643-8. doi: 10.1016/j.biomaterials.2010.01.076. Epub 2010 Feb 9. PMID 20144479
- [Background] Bragdon CR, Greene ME, Freiberg AA, Harris WH, Malchau H. Radiostereometric analysis comparison of wear of highly cross-linked polyethylene against 36- vs 28-mm femoral heads. J Arthroplasty. 2007 Sep;22(6 Suppl 2):125-9. doi: 10.1016/j.arth.2007.03.009. Epub 2007 Jul 26. PMID 17823030
- [Background] Skoldenberg OG, Rysinska AD, Chammout G, Salemyr M, Mukka SS, Boden H, Eisler T. A randomized double-blind noninferiority trial, evaluating migration of a cemented vitamin E-stabilized highly crosslinked component compared with a standard polyethylene component in reverse hybrid total hip arthroplasty. Bone Joint J. 2019 Oct;101-B(10):1192-1198. doi: 10.1302/0301-620X.101B10.BJJ-2019-0456.R2. PMID 31564144
- [Derived] Otten V, Wasterlund D, Lindbjorn J, Mertens C, Mukka S, Crnalic S, Nilsson KG. Evaluation of a new cemented highly cross-linked all-polyethylene cup: a prospective and randomised study assessing wear and fixation characteristics using radiostereometric analysis. Hip Int. 2022 Nov;32(6):779-786. doi: 10.1177/1120700021989991. Epub 2021 Feb 10. PMID 33566703